CLINICAL TRIAL: NCT05510557
Title: The Effect of Blastocyst Morphology and Quality on Obstetric Outcomes in Patients Who Underwent Frozen Embryo Transfer at the Blastocyst Stage: Prospective Cohort Study
Brief Title: Evaluation of Blastocyst Morphology and Quality in Patients With Embryo Transfer at the Blastocyst Stage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, ŞAFAK OLGAN, Associate Professor, Akdeniz University
Other Study IDs: 49849695
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Infertility
Keywords: Embryo Morphology; Frozen - thawed embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective study, the investigators aim to investigate the role of trophectoderm cells and inner cell mass cells on pregnancy outcomes in blastocyst transferred in-vitro fertilization pregnancy. The investigators will support findings with bilateral uterine artery Doppler measurements to be made between the 11th and 14th weeks of pregnancy.

DETAILED DESCRIPTION:
Patients scheduled for thawed blastocyst transfer between May 2022 and December 2022 in Akdeniz University Hospital Center for Reproductive Endocrinology and Assisted Reproduction will be included in the study. Embryos that have reached the Blastocyst stage after the ICSI procedure will be examined by a single experienced embryologist using the ALPHA Istanbul consensus evaluation system.

This system includes separating the blastocyst from the zona pellucida - hatching (Grade 1,2,3,4), the size of ICM and arrangement (grade A, B, C), and the number of TE cells and arrangement (grade A, B, C).

Among the embryos whose quality is determined, the best quality embryo belonging to the patient will be transferred single, patients who develop pregnancy after the transfer will be called for follow-ups for uterine artery Doppler measurements to evaluate uteroplacental flow between 11and 14 weeks, and their Doppler measurements will be recorded. By contacting the patients with the phone numbers recorded at the time of the first visit, the weeks of birth, baby weight, gender, and complications that developed during the pregnancy (Abortion, Preeclampsia, Eclampsia, Fetal Growth Restriction, Oligohydramnios, Polyhydramnios, Gestational Diabetes Mellitus and Antenatal Bleeding) will be recorded.

In case the related relationship can be revealed, the risk situations in terms of complications are determined before the transfer, and it is aimed to increase the number of live births together with the risk-based management in the follow-up and screening programs.

ELIGIBILITY:
Inclusion Criteria:

* Exogenous hormone preparation of the endometrial lining
* Single embryo transfer
* Embryo transfer at the blastocyst stage

Exclusion Criteria:

* Double embryo transfer
* Patients who underwent embryo transfer at the cleavage stage
* >15% loss of embryo viability during embryo thawing
* Patients whose data could not be accessed after follow-up or delivery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients aged 18-40 years who underwent a single freeze-thaw transfer on the 5th day in Akdeniz University Hospital Center for Reproductive Endocrinology and Assisted Reproduction between May 2022 and December 2022 will be included in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Live Birth Rate | 9 months
  pregnancy beyond 24 weeks of gestational age.
Obstetric Complication Rates | 20 weeks after embryo transfer
  Conditions such as preeclampsia, eclampsia, fetal growth restriction, oligohydramnios, polyhydramnios, preterm birth, gestational diabetes mellitus, antenatal bleeding and etc. that develop during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Şafak Olgan, MD, Principal Investigator — 1; Arif C Özsipahi, MD, Study Chair — 2
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)